CLINICAL TRIAL: NCT05044182
Title: Clinical Study of Decompression and Drainage Seton for the Treatment of High Horseshoe Anal Fistula
Brief Title: Decompression and Drainage Seton for Treatment of High Horseshoe Anal Fistula
Acronym: DADS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hui Li, Associate chief physician, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-1-QN-10
Record Dates: First submitted 2021-09-05; First posted 2021-09-14 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula | interventions — Decompression

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decompression and drainage seton (Experimental): Decompress the pressure in intersphincteric space,and drainage seton will be put around the external anal sphincter.
  Interventions: Procedure: Decompression and drainage seton; Procedure: Cutting seton
- Cutting seton (Experimental): Cutting seton will be put around the internal and external anal sphincter.
  Interventions: Procedure: Decompression and drainage seton; Procedure: Cutting seton

INTERVENTIONS:
Procedure: Decompression and drainage seton — Incision the internal sphincter over the fistula tract in intersphinteric space to achieve decompression then drainage seton will be put around external sphincter.
Procedure: Cutting seton — Cutting seton is introduced from outside openning to internal openning and encircling the internal and external anal sphincter.

SUMMARY:
Patients with high horseshoe anal fistula will be randomized to one of two equal group: treatment group will have decompression and drainage seton and control group will undergo cutting seton.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from high horseshoe anal fistula

Exclusion Criteria:

* Specific cause of fistula e.g. Crohn's disease.
* Previous anorectal surgery.
* Patients with malignant tumors or mental illness or other reasons unable to cooperate with the treatment.
* Patients with serious primary diseases such as tumor, malnutrition, endocrine and hematopoietic system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 12 months after the procedure
  recurrence was defined as the clinical reappearance of the fistula after complete healing.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan friendship, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No